CLINICAL TRIAL: NCT00623974
Title: A Phase II Study of Short-Term Use of Teriparatide (Forteo) in the Treatment of Patients With Postoperative Hypocalcemia
Brief Title: Teriparatide (Forteo) in the Treatment of Patients With Postoperative Hypocalcemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0562
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Results first posted 2010-09-13 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Hypocalcemia
Keywords: Hypocalcemia; Teriparatide; Forteo; Calcium; Calcitriol; Rocaltrol
MeSH Terms: conditions — Hypocalcemia | interventions — Teriparatide; Parathyroid Hormone; Calcium; Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Calcium + Calcitriol (Experimental): 1000 milligrams Calcium + 0.25 micrograms Calcitriol orally every 12 hours
  Interventions: Drug: Calcium; Drug: Calcitriol
- Teriparatide 20 mcg (Experimental): Teriparatide at 20 mcg; and 1000 milligrams Calcium + 0.25 micrograms Calcitriol orally every 12 hours
  Interventions: Drug: Teriparatide (Forteo); Drug: Calcium; Drug: Calcitriol
- Teriparatide 40 mcg (Experimental): Teriparatide at 40 mcg; and 1000 milligrams Calcium + 0.25 micrograms Calcitriol orally every 12 hours
  Interventions: Drug: Teriparatide (Forteo); Drug: Calcium; Drug: Calcitriol
- Teriparatide 60 mcg (Experimental): Teriparatide at 60 mcg; and 1000 milligrams Calcium + 0.25 micrograms Calcitriol orally every 12 hours
  Interventions: Drug: Teriparatide (Forteo); Drug: Calcium; Drug: Calcitriol

INTERVENTIONS:
Drug: Teriparatide (Forteo) — Subcutaneous Injection Every 12 Hours for 7 Days
  Other Names: Forteo; PTH; Parathyroid Hormone
  Arms: Teriparatide 20 mcg; Teriparatide 40 mcg; Teriparatide 60 mcg
Drug: Calcium — 1000 milligrams by mouth (PO) Every 12 Hours
Drug: Calcitriol — 0.25 micrograms PO Every 12 Hours
  Other Names: Rocaltrol

SUMMARY:
Primary Objective:

-To identify the optimal dose of a seven-day course of twice-daily teriparatide as compared to standard therapy for hypocalcemia in patients after total thyroidectomy and/or extensive neck dissections (pharyngectomy, laryngectomy,unilateral, bilateral / central neck, mediastinal lymph node neck dissections), with which serum calcium will be raised to corrected serum calcium levels of 8-10.5mg/dL and maintained within this range until the end of the treatment course.

DETAILED DESCRIPTION:
Teriparatide is designed to act like a natural human hormone called parathyroid hormone, which can increase the blood levels of calcium. Calcium plus calcitriol is considered the standard treatment for low calcium in the blood.

After scheduled surgery, the level of calcium in the blood will be monitored according to the standard of care. Between 18 and 24 hours after the surgery, if calcium level drops below an acceptable level, or participants develop symptoms of low calcium, they will be randomly assigned (as in the toss of a coin) to 1 of 4 groups. One group (the "standard-of-care" group) will receive calcium plus calcitriol alone, for 7 days. The other groups (the "teriparatide" groups) will receive 1 of 3 different dose levels of teriparatide for 7 days, plus calcium and calcitriol for 7 days. There is an equal chance of getting assigned to any of these 4 groups, for the first 40 participants enrolled on this study. If enrolled after that point, participants will have a greater chance of being assigned to the group showing the best results.

Standard-of-Care Group:

If assigned to the standard-of-care group, participant will receive calcium and calcitriol according to the standard schedule and dose. The calcium will either be given through a vein or by mouth, and calcitriol will be given by mouth.

Teriparatide Group:

If assigned to a teriparatide group, participant will receive teriparatide by an injection under the skin, twice a day for 7 days. They will be taught how to perform the injections themselves, with a pen-sized device. While in the hospital, the hospital staff will watch them perform the injections and offer help, if needed. If discharged from the hospital and sent home before the 7 days of therapy are complete, they will continue giving themselves the injections (through Day 7) at home. The pen should not be removed from refrigeration for more than 2 -4 hours. Depending on what dose level of teriparatide assigned to receive, they may have to give themselves up to 3 injections each time. In addition to teriparatide, they will receive calcium and calcitriol, according to the standard schedule and dose. The calcium will either be given through a vein or by mouth, and calcitriol by mouth.

Both Groups:

If blood calcium level has not returned to normal after the 7 days of treatment, participants may need to continue receiving calcium and/or calcitriol for as long as the doctor decides it is necessary.

They will be asked to keep a medication log (diary) of when they take the teriparatide and/or calcium/calcitriol. The log should be returned to the research nurse on Day 8.

On Days 1-7, blood will be drawn to check the level of calcium twice a day (while in the hospital) or once a day (while treated as an outpatient). These blood draws (about 1 teaspoon each time) will be performed 2 hours before receiving teriparatide and/or calcium/calcitriol.

Blood will also be drawn to check calcium and parathyroid hormone levels after the study treatment is over. The first of these blood draws (about 1 tablespoon each time) will be performed at 3 days after receiving last dose of teriparatide and/or last dose of calcium/calcitriol. The second blood draw will be performed at 4 weeks after the surgery.

Starting on Day 7, and again at 4 weeks after surgery, they will be asked to collect urine over the course of a 24-hour period so calcium levels can be measured.

From Day 1 to Day 7, if discharged from the hospital and sent home, the study personnel will call on the phone once a day to see how participants are doing. At 3 days after receiving the last dose of teriparatide and/or the last dose of calcium/calcitriol, and at 4 weeks after the surgery, they will be called again.

After the urine collection, blood draw, and phone call at 4 weeks after the surgery, participation in the study is over.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are scheduled for total thyroidectomy, and/or extensive neck dissections (pharyngectomy, laryngectomy, unilateral/bilateral/central neck, and/or mediastinal lymph node neck dissections).
2. Patients who develop, between 18-24 hours after surgery, hypocalcemia as defined by a corrected serum calcium <8.0mg/dL. [Corrected serum calcium (mg/dL) = Measured calcium + (4-albumin) x 0.8]

Exclusion Criteria:

1. Patients who have jejunal tubes
2. Patients <18 years old.
3. Treatment with teriparatide or calcitriol (Rocaltrol) within 1 month prior to surgery
4. Treatment with a bisphosphonate within 3 months prior to surgery
5. Hypercalcemia (corrected serum calcium >10.5mg/dL) or hypocalcemia (corrected serum calcium <8.4mg/dL) on preoperative labs (drawn within 21 days of surgery)
6. Paget's disease of bone
7. Elevated alkaline phosphatase > institutional upper limit of normal (ULN)
8. History of external beam irradiation to the skeleton
9. History of skeletal metastases
10. History of untreated gout
11. History of unstable angina pectoris
12. History of symptomatic orthostatic hypotension
13. Pregnancy (as screened by a serum/urine pregnancy test) or breast-feeding. Female subjects of childbearing potential must have a negative pregnancy test within 7 days of surgery. Postmenopausal women (absence of menses for 12 months) or women with history of hysterectomy or bilateral oophorectomy will not be required to have a pregnancy test. Male and female patients of reproductive potential must agree to utilize an effective form of contraception throughout the study period. The definition of effective contraception will be based on the judgment of the Investigator or designated associate.
14. Hepatic and renal dysfunction defined by the following parameters: (a) Serum AST (SGOT) and ALT (SGPT) > 3 times the institutional ULN, (b) Total serum bilirubin > 2 times the institutional ULN, (c) Serum creatinine > 1.5mg/dL or estimated creatinine clearance < 40mL/min
15. Psychiatric illness or social situation that would limit compliance with study requirements
16. Concomitant use of digoxin
17. Patients may not be receiving any other investigational agents or have participated in any investigational drug study within 28 days preceding the start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mimi Hu, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 2, 2008 to April 13, 2009. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: A total of 7 patients were consented and screened. None of the patients met study entry criteria and thus were not randomized to treatment. Due to slow accrual, the study was closed.
Period: Overall Study
Arm/Group | Calcium + Calcitriol | Teriparatide 20 Mcg | Teriparatide 40 Mcg | Teriparatide 60 Mcg
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcium + Calcitriol | Teriparatide 20 Mcg | Teriparatide 40 Mcg | Teriparatide 60 Mcg | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
Age Continuous [Median (Full Range); unit: years]
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Success
Description: A patient "success" is defined as a normal calcium level (Ca>=8 and Ca<= 10.5) within 48 hours post-treatment initiation and a normal Ca level maintained through day 7 post-treatment initiation.
Time Frame: 2 - 7 days post-treatment
Population: Terminated due low accrual, none of 7 participants met eligibility criteria therefore not treated nor randomized to study arms.
Arm/Group | Calcium + Calcitriol | Teriparatide 20 Mcg | Teriparatide 40 Mcg | Teriparatide 60 Mcg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Study period 1 Year
Description: As no patient received study treatment, neither adverse events nor serious adverse events have occurred.
Arm/Group | Calcium + Calcitriol | Teriparatide 20 Mcg | Teriparatide 40 Mcg | Teriparatide 60 Mcg
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No